CLINICAL TRIAL: NCT05502731
Title: Januse Kinase Inhibition With Filgotinib to Silence Autoreactive B Cells in Rheumatoid Arthritis
Acronym: JAKAR
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Leiden University Medical Center (Other)
Collaborators: Galapagos NV (Industry)
Responsible Party: Principal Investigator, Hans Ulrich Scherer, Associate Professor of Rheumatology, Leiden University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL79681.058.21; 2021-006007-15 (EudraCT Number)
Record Dates: First submitted 2022-08-09; First posted 2022-08-16 (Actual); Last update posted 2022-08-16 (Actual); Status verified 2022-08

CONDITIONS: Rheumatoid Arthritis
Keywords: Autoreactive B cells; Immunological Remission; Anti citrullinated protein antibodies
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — GLPG0634; Adalimumab

STUDY DESIGN:
Intervention Model Description: Open-label, randomized, single center, two-arm, investigator-initiated, interventional clinical study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Add-on filgotinib (Experimental): Treatment with a combination therapy of MTX (7.5 - 15 mg once weekly) and filgotinib p.o. (200 mg once daily) for 24 weeks
  Interventions: Drug: Filgotinib
- Add-on adalimumab (Active Comparator): Treatment with a combination therapy of MTX (7.5 - 15 mg once weekly) and adalimumab s.c. (40 mg biweekly) for 24 weeks
  Interventions: Drug: Adalimumab

INTERVENTIONS:
Drug: Filgotinib — Filgotinib is a small molecule that reversibly inhibits Janus kinases (JAK, selectively JAK 1), thereby inhibiting downstream signalling events induced by various pro-inflammatory and regulatory cytokines.
  Other Names: Jyseleca
  Arms: Add-on filgotinib
Drug: Adalimumab — Adalimumab is a monoclonal antibody selectively inhibiting the pro-inflammatory cytokine TNF-alpha.
  Other Names: Hyrimoz
  Arms: Add-on adalimumab

SUMMARY:
To investigate the effect of filgotinib on phenotype, B cell receptor (BCR) usage and functional parameters of circulating B cells expressing ACPA in patients with ACPA-positive RA that show incomplete response to standard, medium-dose methotrexate (MTX) monotherapy.

DETAILED DESCRIPTION:
B cells expressing anti citrullinated protein antibodies (ACPA) in patients with rheumatoid arthritis (RA) display an activated, proliferative phenotype. Experimental data indicate that ACPA and ACPA-expressing B cells are actively involved in driving the disease process in RA. The present study is based on the hypothesis that targeted intervention with filgotinib as a means to interfere with the activation of B cells in early, active, ACPA-positive RA can reverse the activated, proliferative phenotype of citrullinated antigen-specific B cells.

ELIGIBILITY:
Inclusion Criteria:

Each patient must:

* have a diagnosis of RA and must have fulfilled the revised 2010 EULAR/ACR criteria for classification of RA prior to initiation of first-line treatment.
* have a positive test for the presence of anti-citrullinated protein antibodies (ACPA) in serum with a value of at least 200 U/ml, as determined by routine clinical assay.
* have moderate to highly active disease defined by a disease activity score evaluating 28 joints (DAS28) ≥ 3.2 or, correspondingly, an sDAI score of > 11.
* have used methotrexate monotherapy at a stable, maximally tolerated dose once weekly for at least 3 months; concomitant glucocorticoid therapy is allowed if at a stable dose of ≤ 7.5 mg prednisolon equivalent within 30 days prior to entry in the study.
* have adequate hematologic function (ANC ≥ 4000 cells/μL, platelet count ≥ 150000/μL, and haemoglobin ≥ 10 g/dL (corresponding to 6.2 mmol/L)
* have a serum creatinine clearance of > 15 ml/min.
* be at least 18 years of age
* if female and of childbearing potential, agree to: comply with effective contraceptive measures, use adequate contraception since the last menses and use adequate contraception during the study
* be willing to undergo pre-treatment screening for latent tuberculosis infection by chest X-ray and Mantoux testing as well as serological screening for chronic viral hepatitis infection. As an alternative for the Mantoux test, a standardized IFN-gamma release assay may be used to assess latent tuberculosis infection.
* be able and willing to give written informed consent prior to entry in the study

Exclusion Criteria:

Any patient who:

* has ever been treated with rituximab or another B-cell depleting agent
* has been treated with a biological DMARD (except rituximab) or a targeted synthetic DMARD within 6 months prior to entry in the study
* has received intra-articular or systemic glucocorticoid injections within 30 days prior to baseline or requires narcotic analgesics other than those accepted by the investigator for analgesia (e.g. paracetamol, NSAIDs, codeine, tramadol)
* receives concomitant treatment with a csDMARD other than methotrexate
* has been tested negative for ACPA
* is in clinical remission as defined by a disease activity score evaluating 28 joints (DAS28) ≤ 2.6 or, correspondingly, an sDAI ≤ 3.3
* has evidence of a medical condition which represents a contra-indication for initiation of either a TNF-alpha inhibitor or a Janus kinase inhibitor, as outlined in the SPCs of either adalimumab and/or filgotinib.
* has liver function abnormality (AST and/or ALT ≥ 3 x upper limit of normal range)
* has concurrent treatment with an experimental drug or who has participated in another clinical trial with an investigational drug within 30 days prior to study entry
* has past or current history of solid or haematological neoplasms, except for curatively treated non-melanoma skin cancer, adequately treated in situ carcinoma of the cervix or another cancer curatively treated and with no evidence of disease for at least 10 years
* is pregnant or a currently nursing woman
* is female and of childbearing potential, unwilling to use adequate contraceptive measures during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-10 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Frequency of ACPA-expressing B cells | 24 weeks
  Change from baseline in the frequency of ACPA-expressing B cells secreting ACPA-IgG in ex-vivo PBMC cultures at the 24 week time-point compared between the two treatment arms.

SECONDARY OUTCOMES:
Disease activity | 24 weeks
  Change from baseline in disease activity (assessed as simplified disease activity index (sDAI)) at the 24 week time point. The sDAI is based on an assessment of 28 joints and calculated as the sum of the tender joint count (TJC28), the swollen joint count (SJC28), a patient global assessment on an visual analogue scale (PtGA), an evaluator global assessment (EGA) and the C-reactive Protein level in serum.
Immunological serum/plasma markers | 0, 12, 24 weeks
  Change from baseline in disease- and treatment-related immunological serum/plasma markers (rheumatoid factor (IgM), anti-citrullinated protein antibodies and antibodies against other posttranslational modified proteins (AMPAs), anti-tetanus toxoid antibodies, IgG, IgA, IgM) will be assessed by ELISA and reported as arbitrary units/ml (aU/ml).
B cell receptor (BCR) repertoire | 0, 12, 24 weeks
  Changes to the BCR repertoire of the total circulating B cell pool and of ACPA-expressing B cells at baseline and at the 12 and 24 week time-points using single cell sorting and next generation sequencing.
Secreted ACPA serum repertoire | 0, 12, 24 weeks
  Changes to the secreted ACPA repertoire in serum in relation to the ACPA BCR repertoire using MS-based quantitative antibody clonality screening.
Patient reported outcome parameter: BRAF-MDQ | 0, 12, 24 weeks
  Changes from baseline to the patient reported outcome parameter BRAF-MDQ. The Bristol Rheumatoid Arthritis Fatigue Multidimensional Questionnaire (BRAFMDQ) has been developed to measure broader impacts of rheumatoid arthritis not captured by existing single item PROMs for pain, disability and function. The BRAF-MDQ comprises 20 items (yielding a total score of 0-70) and four subscales of physical fatigue (0-22), living with fatigue (0-21), cognitive fatigue (0-15) and emotional fatigue (0-12), with high scores representing worse fatigue.
Phenotypic cellular markers on circulating lymphocytes | 0, 12, 24 weeks
  Phenotypic cellular markers on circulating lymphocytes (e.g. CD19, CD20, CD27, CD38, CD3, CD4, CD8) will be assessed by flow cytometry and reported as percent expression per cell type.
Patient reported outcome parameter: Netherlands RAID | 0, 12, 24 weeks
  Changes from baseline to the patient reported outcome parameter Netherlands RAID. The Dutch version of the Rheumatoid Arthritis Impact of Disease (RAID) scale is calculated based on 7 Numerical rating scales (NRS) questions. Each NRS is assessed as a number between 0 and 10. The 7 NRS correspond to pain, function, fatigue, sleep, emotional well-being, physical well-being, and coping/self-efficacy. The range of the final RAID value is 0-10 where higher figures indicate worse status.
Patient reported outcome parameter: BRAF-NRS | 0, 12, 24 weeks
  Changes from baseline to the patient reported outcome parameter BRAF-MDQ. The Bristol Rheumatoid Arthritis Numerical Rating Scales (BRAF-NRS) have been developed to measure broader impacts of rheumatoid arthritis not captured by existing single item PROMs for pain, disability and function. The BRAF-NRS comprises three items measuring fatigue severity, effect and coping. The BRAF-NRS for severity and effect have high scores reflecting worse situations (0-10).

CONTACTS AND LOCATIONS:
Overall Officials: Tom WJ Huizinga, MD PhD, Study Chair — Leiden University Medical Center
Locations (1):
- Leiden University Medical Center, Leiden, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
deidentified individual participant data (upon reasonable request)
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Upon publication of the main study results in a scientific journal.

REFERENCES:
- [Background] Kristyanto H, Blomberg NJ, Slot LM, van der Voort EIH, Kerkman PF, Bakker A, Burgers LE, Ten Brinck RM, van der Helm-van Mil AHM, Spits H, Baeten DL, Huizinga TWJ, Toes REM, Scherer HU. Persistently activated, proliferative memory autoreactive B cells promote inflammation in rheumatoid arthritis. Sci Transl Med. 2020 Nov 18;12(570):eaaz5327. doi: 10.1126/scitranslmed.aaz5327. PMID 33208502
- [Background] Kerkman PF, Fabre E, van der Voort EI, Zaldumbide A, Rombouts Y, Rispens T, Wolbink G, Hoeben RC, Spits H, Baeten DL, Huizinga TW, Toes RE, Scherer HU. Identification and characterisation of citrullinated antigen-specific B cells in peripheral blood of patients with rheumatoid arthritis. Ann Rheum Dis. 2016 Jun;75(6):1170-6. doi: 10.1136/annrheumdis-2014-207182. Epub 2015 Jun 1. PMID 26034045
- [Background] Kerkman PF, Rombouts Y, van der Voort EI, Trouw LA, Huizinga TW, Toes RE, Scherer HU. Circulating plasmablasts/plasmacells as a source of anticitrullinated protein antibodies in patients with rheumatoid arthritis. Ann Rheum Dis. 2013 Jul;72(7):1259-63. doi: 10.1136/annrheumdis-2012-202893. Epub 2013 Apr 26. PMID 23625975
- [Background] Scherer HU, Huizinga TWJ, Kronke G, Schett G, Toes REM. The B cell response to citrullinated antigens in the development of rheumatoid arthritis. Nat Rev Rheumatol. 2018 Mar;14(3):157-169. doi: 10.1038/nrrheum.2018.10. Epub 2018 Feb 8. PMID 29416134
- [Background] Westhovens R, Taylor PC, Alten R, Pavlova D, Enriquez-Sosa F, Mazur M, Greenwald M, Van der Aa A, Vanhoutte F, Tasset C, Harrison P. Filgotinib (GLPG0634/GS-6034), an oral JAK1 selective inhibitor, is effective in combination with methotrexate (MTX) in patients with active rheumatoid arthritis and insufficient response to MTX: results from a randomised, dose-finding study (DARWIN 1). Ann Rheum Dis. 2017 Jun;76(6):998-1008. doi: 10.1136/annrheumdis-2016-210104. Epub 2016 Dec 19. PMID 27993829
- [Background] Van Rompaey L, Galien R, van der Aar EM, Clement-Lacroix P, Nelles L, Smets B, Lepescheux L, Christophe T, Conrath K, Vandeghinste N, Vayssiere B, De Vos S, Fletcher S, Brys R, van 't Klooster G, Feyen JH, Menet C. Preclinical characterization of GLPG0634, a selective inhibitor of JAK1, for the treatment of inflammatory diseases. J Immunol. 2013 Oct 1;191(7):3568-77. doi: 10.4049/jimmunol.1201348. Epub 2013 Sep 4. PMID 24006460
- [Background] Hewlett S, Kirwan J, Bode C, Cramp F, Carmona L, Dures E, Englbrecht M, Fransen J, Greenwood R, Hagel S, van de Laar M, Molto A, Nicklin J, Petersson IF, Redondo M, Schett G, Gossec L. The revised Bristol Rheumatoid Arthritis Fatigue measures and the Rheumatoid Arthritis Impact of Disease scale: validation in six countries. Rheumatology (Oxford). 2018 Feb 1;57(2):300-308. doi: 10.1093/rheumatology/kex370. PMID 29087507